CLINICAL TRIAL: NCT02441868
Title: Feasibility Testing of a Hospice Family Caregiver Intervention to Improve Patient Dyspnea Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Margaret Campbell, Professor, Wayne State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDOS-Family
Record Dates: First submitted 2015-04-30; First posted 2015-05-12 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): all participants will receive the training
  Interventions: Behavioral: Shortness of breath recognition and treatment

INTERVENTIONS:
Behavioral: Shortness of breath recognition and treatment — Hospice registered nurses will train family caregivers about how to recognize patient shortness of breath. This training will employ a guided learning tool the Respiratory Distress Observation Scale-Family. Training will be done with a DVD and return demonstration of the skills using the patient. In addition, the family will be taught the bundle of evidence-based interventions to treat shortness of breath.

SUMMARY:
This study is a pilot test of an intervention to train family caregivers of home hospice patients about recognizing and treating shortness of breath.

DETAILED DESCRIPTION:
Shortness of breath is a prevalent symptom causing distress among patients at the end of life. In home hospice care family caregivers are expected to assist their family member with symptom management. This is often accomplished with little or no training.

The investigators have developed a bundle of training materials targeted for family caregivers of home hospice patients at risk for shortness of breath. The investigators will pilot test the intervention in this clinical trial. A future randomized clinical trial is planned and the evidence from this pilot will enhance the planning of that future trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient in home hospice care with an estimated survival of 3-4 weeks, at risk for dyspnea secondary to lung cancer, COPD, or heart failure.
* Family caregiver in patient's home must speak and read English.

Exclusion Criteria:

* Patients with bulbar ALS or quadriplegia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in patient respiratory comfort | Baseline and up to four weeks until patient death
  The Respiratory Distress Observation Scale will be used to measure patient respiratory comfort at enrollment (baseline), twice each week during the study until patient death.

SECONDARY OUTCOMES:
Family caregiver burden index | Baseline and participants will be followed for an average of 4 weeks until date of death
  The Modified Caregiver Strain Index

OTHER OUTCOMES:
Family caregiver stress as measured by Salivary cortisol | Baseline and participants will be followed for an average of four weeks to end at time of death.
  Salivary cortisol
Family anxiety questionnaire | Baseline and participants will be followed for an average of four weeks to end at time of death
  Promis anxiety Short form
Family depression questionnaire | Baseline and participants will be followed for an average of four weeks to end at time of death

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L. Campbell, PhD, Principal Investigator — Wayne State University
Locations (1):
- Angela Hospice, Livonia, Michigan, United States